CLINICAL TRIAL: NCT03270540
Title: Abdominal Ultrasonography in Urinary Tract Infection - When and Why?
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Magdalena Okarska-Napierała, MD, Medical University of Warsaw
Other Study IDs: WarsawMU2W9
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Urinary Tract Infections; UTI
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urinary tract infection (UTI) in a child may be the first symptom of congenital anomaly of the kidneys and the urinary tract (CAKUT). Thus, imaging diagnostics are warranted in children with first episode of UTI.

Abdominal ultrasonography (USG) is the first line imaging modality in evaluating children with UTI. Abnormalities suggesting CAKUT found on USG are an indication for further, more invasive tests. The timing of USG in UTI depends on the clinical situation. It always should be performed urgently when serious acute complications of UTI are suspected. However, appropriate timing of USG in children responding well to therapy, is a matter of debate. According to animal studies, E. coli produces toxin which dilates the urinary tract. This may result in misleading picture on USG in acute phase of infection. Guidelines on UTI management in children differ in respect to recommended USG timing.

The purpose of the study is to investigate how UTI does affect USG results in children and when its effect subsides.

Methods 150 children up to 3 years of age, with the first episode of UTI, will be included in our study. Three USG examinations will be performed by single radiologist in every child:

1. in the first day of treatment,
2. two weeks after treatment initiation,
3. four weeks after treatment initiation. Age, gender, etiologic factor, C-reactive protein concentration and white blood cells count will be included in statistical analysis.

The study is aimed to help clinicians interpret USG findings during UTI and make reasonable plans for further imaging diagnostics in children with UTI.

ELIGIBILITY:
Inclusion Criteria:

- laboratory diagnosis of UTI in a child (positive leucocyturia and significant bacteriuria)

Exclusion Criteria:

* known previous UTIs
* known congenital abnormality of the kidney and the urinary tract (CAKUT)

Max Age: 3 Years | Sex: All
Age Groups: Child
Study Population: children with UTI treated in Medical University of Warsaw Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-11-18 (Actual); Study Completion 2018-11-18 (Actual)

PRIMARY OUTCOMES:
USG abnormality persistence | 4 weeks
  significant abnormalities within kidney size or calices/pelvis/ureter dimensions, reproducible in subsequent USG examinations

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw Children's Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: National Institute for Health and Care Excellence. Urinary tract infections in children and young people 2013 July — https://www.nice.org.uk/guidance/qs36
- See also: European Association of Urology; European Society for Pediatric Urology Urinary tract infections in children: (EAU/ESPU) guidelines. — http://uroweb.org/guideline/paediatric-urology/#3
- See also: Canadian Paediatric Society, Urinary tract infection in infants and children: Diagnosis and management — http://www.cps.ca/en/documents/position/urinary-tract-infections-in-children